CLINICAL TRIAL: NCT03754959
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 1358894 (Double-blind, Randomised, Placebo-controlled, Parallel-group Design) and Evaluation of Midazolam Interaction (Nested, Open, Fixed-sequence, Intra-individual Comparison) in Healthy Male Subjects
Brief Title: This Study in Healthy Men Tests How Different Doses of BI 1358894 Are Taken up in the Body and How Well They Are Tolerated. The Study Also Tests How BI 1358894 Affects the Way the Body Breaks Down Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1402-0002; 2018-000389-12 (EudraCT Number)
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Group 1 (Experimental)
  Interventions: Drug: BI 1358894; Drug: Placebo; Drug: Midazolam
- Dose Group 2 (Experimental)
  Interventions: Drug: BI 1358894; Drug: Placebo; Drug: Midazolam
- Dose Group 3 (Experimental)
  Interventions: Drug: BI 1358894; Drug: Placebo; Drug: Midazolam
- Dose Group 4 (Experimental)
  Interventions: Drug: BI 1358894; Drug: Placebo; Drug: Midazolam
- Dose Group 5 (Experimental)
  Interventions: Drug: BI 1358894; Drug: Placebo; Drug: Midazolam

INTERVENTIONS:
Drug: BI 1358894 — Film-coated tablet
Drug: Placebo — Film-coated tablet
Drug: Midazolam — Solution for injection

SUMMARY:
The primary objective of the trial is to investigate the safety and tolerability of BI 1358894 in healthy male subjects following oral administration of multiple rising doses over 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use adequate contraception with their female partner throughout the study and until one month after the last administration of trial medication. Adequate methods are:

  * Sexual abstinence or
  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide) Unprotected sexual intercourse with a female partner is not allowed throughout the study and until one month after the last administration of trial medication.

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* C-Reactive Protein > upper limit of normal (ULN), erythrocyte sedimentation rate (ESR) ≥15 millimeters/h, liver or kidney parameter above ULN, or any other laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Positive or missing faecal occult blood test (retest allowed)
* Positive testing for faecal calprotectin (retest allowed)
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during in-house confinement
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

REFERENCES:
- [Derived] Fuertig R, Goettel M, Herich L, Hoefler J, Wiebe ST, Sharma V. Effects of Single and Multiple Ascending Doses of BI 1358894 in Healthy Male Volunteers on Safety, Tolerability and Pharmacokinetics: Two Phase I Partially Randomised Studies. CNS Drugs. 2023 Dec;37(12):1081-1097. doi: 10.1007/s40263-023-01041-4. Epub 2023 Nov 29. PMID 38019355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety, tolerability, and pharmacokinetics of multiple rising oral doses of BI 1358894 (double-blind, randomised, placebo-controlled, parallel-group design) and evaluation of midazolam interaction (nested, open, fixed-sequence, intra-individual comparison) in healthy male subjects
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they met all implemented inclusion/exclusion criteria, Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated
Groups:
- Placebo Matching BI 1358894 Dose Group: Oral administration of placebo matching to BI 1358894 film-coated tablet with 240 milliliter (mL) of water after a standard continental breakfast once per day from day 1 to day 14
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 Placebo matching to BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 10 Milligram (mg) Dose Group: Oral administration of 10 milligram (mg) BI 1358894 film-coated tablet (2*5 mg tablet) once daily for 14 days with 240 milliliter (mL) water after a standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 25 Milligram (mg) Dose Group: Oral administration of 25 milligram (mg) BI 1358894 film-coated tablet (1*25 mg tablet) once daily for 14 days with 240 milliliter (mL) water after a standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 50 Milligram (mg) Dose Group: Oral administration of 50 milligram (mg) BI 1358894 film-coated tablet (2*25 mg tablet) once daily for 14 days with 240 milliliter (mL) water after standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 100 Milligram (mg) Dose Group: Oral administration of 100 milligram (mg) BI 1358894 film-coated tablet (1*100 mg tablet) once daily for 14 days with 240 milliliter (mL) water after standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 200 Milligram (mg) Dose Group: Oral administration of 200 milligram (mg) BI 1358894 film-coated tablet (2*100 mg tablet) once daily for 14 days with 240 milliliter (mL) water after standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
Period: Overall Study
Arm/Group | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Started | 10 | 8 | 8 | 8 | 8 | 8
Completed | 10 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who received at least one dose of study drug. This was the full analysis set population in the sense of ICH-E9. It was used for analysis of safety (except for the ECG exposure-response analyses), demographic data, and baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group | Total
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.1 (9.7) | 32.0 (8.1) | 32.4 (6.8) | 32.3 (7.7) | 29.3 (1.8) | 26.3 (5.1) | 30.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 8 | 8 | 8 | 8 | 8 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 8 | 8 | 8 | 6 | 8 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 10 | 8 | 7 | 8 | 8 | 8 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With On-treatment Drug-related Adverse Events (AEs).
Description: Number of subjects with on-treatment drug-related Adverse Events (AEs).
Time Frame: Midazolam: Up to 1 day, BI 1358894 or Placebo + Midazolam: Up to 1 day and BI 1358894: Up to 13 days.
Population: Treated set (TS): all subjects who received at least one dose of study drug. This was the full analysis set population in the sense of ICH-E9.
Measure: Number; unit: Participants
Groups:
- Midazolam: Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL with 240 milliliter (mL) water after a standard continental breakfast on Day -1 before administration of BI 1358894/ Placebo
- Placebo + Midazolam: Oral administration of placebo matching to BI 1358894 film-coated tablet with 240 milliliter (mL) of water after a standard continental breakfast once per day from day 1 to day 14.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 placebo matching to BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 10 mg + Midazolam; BI 1358894 10 Milligram (mg) Dose Group: Oral administration of 10 milligram (mg) BI 1358894 film-coated tablet (2*5 mg tablet) once daily for 14 days with 240 milliliter (mL) water after a standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 25 mg + Midazolam: Oral administration of 25 milligram (mg) BI 1358894 film-coated tablet (1*25 mg tablet) once daily for 14 days with 240 milliliter (mL) water after a standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894was administered immediately prior to midazolam.
- BI 1358894 50 mg + Midazolam; BI 1358894 50 Milligram (mg) Dose Group: Oral administration of 50 milligram (mg) BI 1358894 film-coated tablet (2*25 mg tablet) once daily for 14 days with 240 milliliter (mL) water after standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 100 mg + Midazolam; BI 1358894 100 Milligram (mg) Dose Group: Oral administration of 100 milligram (mg) BI 1358894 film-coated tablet (1*100 mg tablet) once daily for 14 days with 240 milliliter (mL) water after standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- BI 1358894 200 mg + Midazolam: Oral administration of 200 milligram (mg) BI 1358894 film-coated tablet (2*100 mg tablet) once daily for 14 days with 240 milliliter (mL) water after standard continental breakfast.
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
- Placebo Matching BI 1358894 Dose Group: Oral administration of placebo matching to BI 1358894 film-coated tablet with 240 milliliter (mL) of water after a standard continental breakfast once per day from day 1 to day 14
  Oral administration of midazolam as solution for injection (5 mg/5 mL) diluted to 50 microgram (μg)/mL*1.5 mL (75 μg) with 240 milliliter (mL) water as three single doses on days -1, 1 and 14, after a standard continental breakfast.
  On Day 1 and 14 BI 1358894 was administered immediately prior to midazolam.
Arm/Group | Midazolam | Placebo + Midazolam | BI 1358894 10 mg + Midazolam | BI 1358894 25 mg + Midazolam | BI 1358894 50 mg + Midazolam | BI 1358894 100 mg + Midazolam | BI 1358894 200 mg + Midazolam | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 50 | 10 | 8 | 8 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 8 | 8
Participants | 0 | 1 | 4 | 4 | 3 | 4 | 5 | 6 | 2 | 5 | 1 | 4 | 5

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma Over a Time Interval 0 to 24 h After Administration of the First Dose
Description: Area under the concentration-time curve of the analyte in plasma over a time interval 0 to 24 hours (h) after administration of the first dose (AUC0-24).
Time Frame: Within 2 hours before and 0.17, 0.33, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 27, 48, 72, 75, 96, 120, 123, 144, 192, 195, 240, 243, 288, 311, 312.17, 312.33, 312.5, 313, 314, 315, 316, 318, 320, 324, 336, 360, 384, 408, 432, 456, 504 hours after administration.
Population: Pharmacokinetic parameter set (PKS): all subjects in the TS who provided at least 1 PK parameter that was not excluded due to a protocol deviation relevant to the statistical evaluation of PK endpoints or due to PK non-evaluability, only subjects with available data were included in the endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomols * hours per liter
Arm/Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 8 | 8 | 6 | 8 | 8
nanomols * hours per liter | 801 (22.7) | 1570 (28.0) | 2690 (17.5) | 5520 (18.3) | 8200 (13.3)

3. Secondary Outcome: Maximum Measured Concentration of BI 1358894 in Plasma
Description: Maximum measured concentration of the analyte BI 1358894 in plasma (Cmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol per liter
Arm/Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8
Nanomol per liter | 78.8 (16.0) | 152 (34.7) | 217 (28.3) | 491 (17.2) | 634 (20.8)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 1358894 in Plasma at Steady State Over a Uniform Dosing Interval τ
Description: Area under the concentration-time curve of BI 1358894 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol * hours per liter
Arm/Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
nanomol * hours per liter | 2070 (27.1) | 3520 (27.8) | 5890 (35.1) | 12600 (16.3) | 18900 (13.5)

5. Secondary Outcome: Maximum Measured Concentration of BI 1358894 in Plasma at Steady State Over a Uniform Dosing Interval τ
Description: Maximum measured concentration of BI 1358894 in plasma at steady state over a uniform dosing interval τ (Cmax,ss)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol per liter
Arm/Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
nanomol per liter | 138 (14.5) | 225 (18.8) | 383 (26.7) | 843 (19.8) | 1150 (13.8)

6. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (Day 1)
Description: Area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: 25.5, 23.83, 23.5, 23, 22, 21.5, 21, 20, 18, 16 and 1 hour before and 0.17, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 311, 312.33, 312.5, 313, 314, 314.5, 315, 316, 318 and 320 hours after administration of BI 1358894 .
Population: PKS-Midazolam (PKS-MDZ): all subjects from the TS receiving BI 1358894 or placebo and midazolam who provided at least one secondary PK parameter for midazolam that was not excluded according to the description above. It was used for investigation of relative bioavailability
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomol * hours per liter
Arm/Group | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8
picomol * hours per liter
  Midazolam + BI 1358894 or Placebo | 2960 (31.8) | 3630 (47.2) | 3120 (29.6) | 2810 (37.2) | 3360 (26.3) | 2480 (24.1)
  Midazolam | 3030 (28.6) | 3790 (46.0) | 3090 (28.6) | 3000 (40.2) | 3610 (22.1) | 2750 (28.2)
Statistical Analysis 1: Comparison: Placebo Matching BI 1358894 Dose Group; The statistical model used for the analysis of the secondary endpoints was an ANOVA model on the logarithmic scale including 'treatment' ('midazolam' and 'midazolam + Placebo/BI') as fixed effect and 'subject' as random effect. The analysis was performed separately for Day 1 and Day 14; Test type: Other; Ratio = 97.9, 90% CI 2-sided [90.2 to 106.2] — Ratio is calculated with Placebo+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 2: Comparison: BI 1358894 10 Milligram (mg) Dose Group; Test type: Other; Ratio = 95.9, 90% CI 2-sided [89.9 to 102.4] — Ratio is calculated with BI 1358894 10 mg+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 3: Comparison: BI 1358894 25 Milligram (mg) Dose Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 101.0, 90% CI 2-sided [96.3 to 106.1] — Ratio is calculated with BI 1358894 25 mg+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 4: Comparison: BI 1358894 50 Milligram (mg) Dose Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 93.7, 90% CI 2-sided [86.8 to 101.1] — Ratio is calculated with BI 1358894 50 mg+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 5: Comparison: BI 1358894 100 Milligram (mg) Dose Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 93.1, 90% CI 2-sided [87.3 to 99.3] — Ratio is calculated with BI 1358894 100 mg+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 6: Comparison: BI 1358894 200 Milligram (mg) Dose Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 90.0, 90% CI 2-sided [83.8 to 96.7] — Ratio is calculated with BI 1358894 200 mg+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator

7. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (Day 14)
Description: as for outcome 6
Time Frame: 25.5, 23.83, 23.5, 23, 22, 21.5, 21, 20, 18, 16 and 1 hour before and 0.17, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 311, 312.33, 312.5, 313, 314, 314.5, 315, 316, 318 and 320 hours after administration of BI 1358894.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomol * hours per liter
Arm/Group | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 mg + Midazolam | BI 1358894 50 mg + Midazolam | BI 1358894 100 mg + Midazolam | BI 1358894 200 mg + Midazolam
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8
picomol * hours per liter
  Midazolam + BI 1358894 or Placebo: number analyzed (Participants) | 10 | 8 | 7 | 7 | 8 | 8
  Midazolam + BI 1358894 or Placebo | 3200 (28.9) | 4450 (43.3) | 3360 (26.0) | 3440 (17.3) | 3480 (23.6) | 2460 (23.4)
  Midazolam | 3030 (28.6) | 3790 (46.0) | 3090 (28.6) | 3000 (40.2) | 3610 (22.1) | 2750 (28.2)
Statistical Analysis 1: Comparison: Placebo Matching BI 1358894 Dose Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 105.7, 90% CI 2-sided [95.6 to 116.9] — Ratio is calculated with Placebo+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 2: Comparison: BI 1358894 10 Milligram (mg) Dose Group; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 117.5, 90% CI 2-sided [106.5 to 129.6] — Ratio is calculated with BI 1358894 10 mg+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 3: Comparison: BI 1358894 25 mg + Midazolam; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 112.6, 90% CI 2-sided [102.9 to 123.1] — Ratio is calculated with BI 1358894 25 mg+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 4: Comparison: BI 1358894 50 mg + Midazolam; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 110.3, 90% CI 2-sided [90.1 to 135.1] — Ratio is calculated with BI 1358894 50 mg+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 5: Comparison: BI 1358894 100 mg + Midazolam; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 96.4, 90% CI 2-sided [84.5 to 110.1] — Ratio is calculated with BI 1358894 100 mg+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 6: Comparison: BI 1358894 200 mg + Midazolam; [analysis description as in outcome 6, analysis 1]; Test type: Other; Ratio = 89.3, 90% CI 2-sided [74.9 to 106.4] — Ratio is calculated with BI 1358894 200 mg+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator

8. Secondary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Day 1)
Description: Maximum measured concentration of midazolam in plasma (Cmax).
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole per liter
Arm/Group | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8
picomole per liter
  Midazolam + BI 1358894 or placeobo (T) | 913 (26.2) | 1090 (32.1) | 1130 (30.5) | 920 (32.8) | 1150 (19.0) | 812 (19.7)
  Midazolam (R) | 929 (25.6) | 1120 (34.1) | 963 (42.0) | 974 (35.0) | 1170 (8.89) | 828 (30.6)
Statistical Analysis 1: Comparison: Placebo Matching BI 1358894 Dose Group; The statistical model used for the analysis of the secondary endpoints was an ANOVA mode lon the logarithmic scale including 'treatment' ('midazolam' and 'midazolam + Placebo/BI') as fixed effect and 'subject' as random effect. The analysis was performed separately for Day 1 and Day 14; Test type: Other; Ratio = 98.3, 90% CI 2-sided [84.2 to 114.8] — Ratio is calculated with Placebo+Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 2: Comparison: BI 1358894 10 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 98.0, 90% CI 2-sided [87.9 to 109.3] — Ratio is calculated with BI 1358894 10mg +Midazolam on day 1 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 3: Comparison: BI 1358894 25 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 117.5, 90% CI 2-sided [102.6 to 134.6] — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 4: Comparison: BI 1358894 50 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 94.5, 90% CI 2-sided [85.5 to 104.4] — [estimate comment as in outcome 6, analysis 4]
Statistical Analysis 5: Comparison: BI 1358894 100 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 98.2, 90% CI 2-sided [87.3 to 99.3] — [estimate comment as in outcome 6, analysis 5]
Statistical Analysis 6: Comparison: BI 1358894 200 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 98.0, 90% CI 2-sided [84.3 to 114.0] — [estimate comment as in outcome 6, analysis 6]

9. Secondary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Day 14)
Description: Maximum measured concentration of midazolam in plasma (Cmax).
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole per liter
Arm/Group | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8
picomole per liter
  Midazolam + BI 1358894 or placeobo (T): number analyzed (Participants) | 10 | 8 | 7 | 7 | 8 | 8
  Midazolam + BI 1358894 or placeobo (T) | 887 (27.1) | 1180 (28.2) | 1070 (31.0) | 1090 (27.3) | 985 (29.3) | 722 (18.8)
  Midazolam (R) | 929 (25.6) | 1120 (34.1) | 963 (42.0) | 974 (35.0) | 1170 (8.89) | 828 (30.6)
Statistical Analysis 1: Comparison: Placebo Matching BI 1358894 Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 95.5, 90% CI 2-sided [81.3 to 112.1] — Ratio is calculated with Placebo+Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 2: Comparison: BI 1358894 10 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 105.7, 90% CI 2-sided [91.5 to 122.0] — Ratio is calculated with BI 1358894 10mg +Midazolam on day 14 in the nominator and the Midazolam on day -1 in the denominator
Statistical Analysis 3: Comparison: BI 1358894 25 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 116.3, 90% CI 2-sided [90.9 to 148.7] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 4: Comparison: BI 1358894 50 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 106.8, 90% CI 2-sided [92.4 to 123.4] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 5: Comparison: BI 1358894 100 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 83.9, 90% CI 2-sided [71.2 to 98.9] — [estimate comment as in outcome 7, analysis 5]
Statistical Analysis 6: Comparison: BI 1358894 200 Milligram (mg) Dose Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; Ratio = 87.2, 90% CI 2-sided [73.5 to 103.5] — [estimate comment as in outcome 7, analysis 6]

ADVERSE EVENTS:
Time Frame: Midazolam AE collection: Up to 1 day BI 1358894 or Placebo + Midazolam AE collection: Up to 1 day BI 1358894 AE collection: Up to 13 days All-cause mortality: Up to 17 days
Description: Treated set (TS): all subjects who received at least one dose of study drug.
Arm/Group | Midazolam | Placebo + Midazolam | BI 1358894 10 mg + Midazolam | BI 1358894 25 mg + Midazolam | BI 1358894 50 mg + Midazolam | BI 1358894 100 mg + Midazolam | BI 1358894 200 mg + Midazolam | Placebo Matching BI 1358894 Dose Group | BI 1358894 10 Milligram (mg) Dose Group | BI 1358894 25 Milligram (mg) Dose Group | BI 1358894 50 Milligram (mg) Dose Group | BI 1358894 100 Milligram (mg) Dose Group | BI 1358894 200 Milligram (mg) Dose Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/50 | 1/10 | 4/8 | 4/8 | 3/8 | 4/8 | 5/8 | 7/10 | 3/8 | 6/8 | 1/8 | 4/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam (N=50) | Placebo + Midazolam (N=10) | BI 1358894 10 mg + Midazolam (N=8) | BI 1358894 25 mg + Midazolam (N=8) | BI 1358894 50 mg + Midazolam (N=8) | BI 1358894 100 mg + Midazolam (N=8) | BI 1358894 200 mg + Midazolam (N=8) | Placebo Matching BI 1358894 Dose Group (N=10) | BI 1358894 10 Milligram (mg) Dose Group (N=8) | BI 1358894 25 Milligram (mg) Dose Group (N=8) | BI 1358894 50 Milligram (mg) Dose Group (N=8) | BI 1358894 100 Milligram (mg) Dose Group (N=8) | BI 1358894 200 Milligram (mg) Dose Group (N=8)
Headache (Nervous system disorders) | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 4 | 0 | 5 | 1 | 1 | 5
Orthostatic intolerance (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03754959/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT03754959/SAP_001.pdf